CLINICAL TRIAL: NCT01525771
Title: A Phase I-II Study of Systemic Capecitabine, Cisplatin and Intraperitoneal Docetaxel (XPID) in Patients With Advanced Stomach Cancer With Peritoneal Seeding
Brief Title: Safety Study of Combined Systemic and Intraperitoneal Chemotherapy to Treat Stomach Cancer
Acronym: XPID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-XPID-1
Record Dates: First submitted 2011-07-18; First posted 2012-02-03 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Stage IV Gastric Cancer With Metastasis
Keywords: Advanced Gastric cancer; Xeloda (Capecitabine); Cisplatin; Taxotere (Docetaxel)
MeSH Terms: interventions — Docetaxel; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No intervention (No Intervention): Single-center, open-label, prospective, single-arm, phase I-II study
  Interventions: Other: Docetaxel

INTERVENTIONS:
Other: Docetaxel — The study medication will be administered every 3 weeks for a maximum of 8cycles. A study medication will be given to the patients.
  * Docetaxel (-1 to 3 level)mg/m2 IV(D1) every 21 days (-1 level: 40, 1 level: 60, 2 level: 80, 3 level: 100)
  * Xeloda 937.5 mg/m2/ day PO, twice a day(D1-D14) every 21 days
  * Cisplatin 60mg/m2 IV (D1) every 21 days
  Other Names: XP with Intraperitoneal Docetaxel; Capecitabine; Cisplatin

SUMMARY:
A maximum of 8 cycles of chemotherapy will be administered. Depending on patients' tolerability, 8 cycles of chemotherapy will be given to the patients.

DETAILED DESCRIPTION:
Single-center, open-label, prospective, single-arm, phase I-II study

About 37 patients (Phase I 18, Phase II 31 (including 12 patients from Phase I)

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable or metastatic advanced gastric adenocarcinoma confirmed by histology
2. Peritoneal seeding proven by histology or cytology
3. Completion of adjuvant chemotherapy 6 months before the study, or no previous chemotherapy (But, patients who received docetaxel or cisplatin as adjuvant chemotherapy should be excluded)
4. Age 18 to 70 years old
5. Eastern Cooperative Oncology Group performance status <_ 2
6. Estimated life expectancy of more than 3 months
7. Adequate bone marrow function (WBCs>3,000/µL and absolute neutrophil count (ANC) >1,500/µL and platelets>100,000/µL),
8. Adequate renal function: creatinine < 1 x upper normal limit (UNL) or creatinine clearance _> 60ml/min
9. Adequate hepatic function: bilirubin < 1.5 x UNL, AST/ALT levels < 2.5 x UNL, alkaline phosphatase < 5 x UNL (except in case of bone metastasis without any liver disease)
10. Written informed consent

Exclusion Criteria:

1. Contraindication to any drug contained in the chemotherapy regimen
2. Other tumor type than adenocarcinoma
3. Presence or history of CNS metastasis
4. Gastric outlet or bowel obstruction
5. Evidence of serious gastrointestinal bleeding
6. Peripheral neuropathy > grade 2
7. History of significant neurologic or psychiatric disorders
8. History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
9. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
10. Other serious illness or medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  Phase I Study
  - Maximum tolerated dose of Intraperitoneal Docetaxel
  Phase II Study
  * Progression-free survival rate at 6 months
  * response rate, time to progression, overall survival

SECONDARY OUTCOMES:
Safety profile | 1 year
Overall survival | 1 year
Progression free survival | 1 year
efficacy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, MD, Principal Investigator — Asan Medical Center/Univ of Ulsan
Locations (1):
- Asan Medical Center, Seoul, South Korea